CLINICAL TRIAL: NCT01704001
Title: A Post-Marketing Clinical Pharmacokinetics Study of ART-123 in DIC Subjects With Renal Impairment
Brief Title: Clinical Pharmacokinetics Study of ART-123 in Disseminated Intravascular Coagulation (DIC) Subjects With Renal Impairment
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Asahi Kasei Pharma Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ART-123 IV-2
Record Dates: First submitted 2012-10-01; First posted 2012-10-11 (Estimated); Last update posted 2017-02-15 (Actual); Status verified 2012-10

CONDITIONS: Disseminated Intravascular Coagulation
Keywords: ART-123; Disseminated Intravascular Coagulation; Pharmacokinetics
MeSH Terms: conditions — Disseminated Intravascular Coagulation | interventions — ART123

ARMS (4):
- Renal impairment grade 0 (Experimental)
  Interventions: Drug: ART-123
- Renal impairment grade 1 (Experimental)
  Interventions: Drug: ART-123
- Renal impairment grade 2 (Experimental)
  Interventions: Drug: ART-123
- Renal impairment grade 3 (Experimental)
  Interventions: Drug: ART-123

INTERVENTIONS:
Drug: ART-123 — 380 U/kg/day or 130 U/kg/day(Subjects with severe renal impairment) for 6 days
  Other Names: Recomodulin™

SUMMARY:
To investigate the impact of impaired renal function on the pharmacokinetics of ART-123 in patients with Disseminated Intravascular Coagulation.

To investigate the safety of ART-123 in patients with Disseminated Intravascular Coagulation.

ELIGIBILITY:
Inclusion Criteria:

* Japanese Association for Acute Medicine-defined DIC criteria score >= 4
* Written informed consent from patient or guardian

Exclusion Criteria:

* Patients showing intracranial, pulmonary, gastrointestinal hemorrhage
* Patients with a history of cerebrovascular disorders within the past 52 week
* Patients with a history of hypersensitivity to the ingredients of ART-123 preparations
* Pregnant women, nursing mothers or possibly pregnant women

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2012-10; Primary Completion 2013-10 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Composite of Pharmacokinetics | pre-dose, 0,2,4,8,24 hours post-dose
  Cmax, Area Under Curve, T1/2,CLtot,CLR
Incidence rate of hemorrhage related adverse events | from the start of infusion to 8days after the cessation of infusion

CONTACTS AND LOCATIONS:
Locations (1):
- Ōita, Japan